CLINICAL TRIAL: NCT05969366
Title: Early Clinical and Radiological Outcomes of Uncemented Fully Coated Stem With Patients of 85 Years and More, Complications and Risks Factor
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Olivier ROCHE, Praticien Hospitalier, Central Hospital, Nancy, France
Other Study IDs: 2022PI032
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Arthroplasty Complications
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients 85 yearsold or orlder who hab total hip replacement with uncemented femoral stem
  Interventions: Procedure: Total hip arthroplasty

INTERVENTIONS:
Procedure: Total hip arthroplasty

SUMMARY:
Retrospective, single-centre study. Review of patients aged 85 and over who underwent total hip replacement between June 2015 and February 2022.

This is a femoral stem survival study with calculation of the complication rate in this population.

The study does not focus on total hip replacements in the context of trauma. The secondary endpoint was the search for complication risk factors.

ELIGIBILITY:
Inclusion Criteria:

* receive total hip arthroplasty with uncemented stem fully hydroxyapatites coated

Exclusion Criteria:

* trauma context
* less than 3 month follow up
* Any surgery of the hip as medical history

Min Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Any people of 85 years of more who received total hip arthroplasty with uncemented stem fully hydroxyapatitis coated
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2023-07 (Actual)

PRIMARY OUTCOMES:
rate of complication | minimum of 3 months follow up
  survival study, any complications

SECONDARY OUTCOMES:
risk factor of complications | minimum of 3 months follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Emile Gallé, Nancy, France